CLINICAL TRIAL: NCT07127627
Title: Characterization of Abdomino-pelvic Lesions in Cancer Patients by 18F-FDG PET/CT
Brief Title: Characterization of Abdomino-pelvic Lesions by 18Fluorine- Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography
Acronym: 18F-FDG PET/CT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma A samy, assistant lecturer of nuclear medicine, Assiut University
Other Study IDs: characterization by PET/CT
Record Dates: First submitted 2025-08-09; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Abdominal Sepsis
Keywords: abdominopelvic lesions
MeSH Terms: conditions — Intraabdominal Infections | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PET/CT — positron emission tomography/computed tomography

SUMMARY:
The aim of the study is to identify and characterize lesions in the abdominopelvic region detected by 18fluorine- fluorodeoxyglucose (FDG) positron Emission Tomography combined Computed Tomography (PET/CT) scan, including determining their malignant or benign nature, and to determine the extent of disease to facilitate proper management

DETAILED DESCRIPTION:
positron Emission Tomography combined Computed Tomography is a hybrid imaging that provides both anatomical and functional data that helps to differentiate between benign and malignant diseases. [18F]FDG is taken up by both normal cells utilizing glucose like (kidneys, ureters and urinary bladder due to urinary excretion, Variable degrees of uptake can also seen in the liver, spleen, bone marrow, bowel, testes and uterus) .and also the tumor cells which usually have a high glucose demand. This uptake is mediated by the cell surface carrier molecules designated as glucose transporters (GLUT) and can be measured with the semi quantitative index called standardized uptake values (SUV) Cancer cells divide rapidly and have greater metabolic rates. Through the upregulation of glucose transport proteins on the cell membrane, cancer cells exhibit enhanced glucose uptake . Studies have demonstrated that SUV of 2.5 can differentiate malignant versus benign tissues , thus, Proper characterization of abdomino-pelvic lesions will lead to improve chances for successful management and treatment.

Multiple studies have shown that Dual-time point (DTP) 18F-FDG PET/CT may provide more help in the differentiation of malignant lesions from benign ones.as Dual-Time-Point PET/CT involves two scans, one early and one delayed, allowing for the assessment of FDG uptake kinetics, malignant tumors tend to show increased FDG uptake over time, indicating higher glucose metabolism. But benign Lesions or those with inflammatory processes may show a decrease or no significant change in FDG uptake over time.

FDG activity in urine interferes with tumor activity. Therefore, the value of FDG PET has only a limited role in detecting tumors in the bladder wall and urinary tract, Thus several methods have been investigated and tested to reduce urine FDG activity: catheterization, dual-phase imaging, early PET images, late PET images after voiding, oral hydration, and forced diuresis

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: All of the patients were suspected of having malignancy (new, recurrent or metastatic) based on pathology or conventional radiological studies and were referred to nuclear medicine unit for 18F-FDG-PET-CT scan

Exclusion Criteria:

* patients underwent recent abdominal or pelvic surgery.
* patients with blood glucose level ˃200 mg/dL
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients were suspected of having malignancy (new, recurrent or metastatic) based on pathology or conventional radiological studies and were referred to nuclear medicine unit for 18F-FDG-PET-CT scan
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of 18F FDG PET/CT | 3 years
  identify and characterize abdominopelvic lesions, initial staging, follow up of treatment and detection of recurrence in the abdominopelvic region, including determining their malignant or benign nature, and to determine the extent of disease, Assess the spread of disease to lymph nodes, distant metastases, or other areas, to facilitate proper management.

SECONDARY OUTCOMES:
Evaluate the diagnostic power of alternative technologies | 3 years
  Evaluate the diagnostic power of alternative technologies like dual time point images, bladder evacuation and forced diuresis in characterizing abdominopelvic lesions.

REFERENCES:
- [Background] Bouchelouche K. PET/CT in Bladder Cancer: An Update. Semin Nucl Med. 2022 Jul;52(4):475-485. doi: 10.1053/j.semnuclmed.2021.12.004. Epub 2022 Jan 5. PMID 34996595
- [Background] Khandelwal Y, Singh Parihar A, Sistani G, Ramirez-Fort MK, Zukotynski K, Subramaniam RM. Role of PET/Computed Tomography in Gastric and Colorectal Malignancies. PET Clin. 2024 Apr;19(2):177-186. doi: 10.1016/j.cpet.2023.12.004. Epub 2024 Jan 9. PMID 38199915
- [Background] Wang J, Liu X. Medical image recognition and segmentation of pathological slices of gastric cancer based on Deeplab v3+ neural network. Comput Methods Programs Biomed. 2021 Aug;207:106210. doi: 10.1016/j.cmpb.2021.106210. Epub 2021 May 29. PMID 34130088
- [Background] Sartin SL, Shetty DR, Strange CD, Gayer G, Ahuja J, Agrawal R, Truong MT. Pitfalls in Positron Emission Tomography/Computed Tomography in the Thorax and Abdomen. Semin Ultrasound CT MR. 2024 Dec;45(6):488-495. doi: 10.1053/j.sult.2024.07.012. Epub 2024 Jul 26. PMID 39069275
- [Background] Cao Y, Zhou K, Diao W, Long X, Tian F, Su M, Jia Z. Age-related changes of standardized uptake values in the blood pool and liver: a decade-long retrospective study of the outcomes of 2,526 subjects. Quant Imaging Med Surg. 2021 Jan;11(1):95-106. doi: 10.21037/qims-20-35. PMID 33392014